CLINICAL TRIAL: NCT03829033
Title: Photon Therapy Versus Proton Therapy in Early Tonsil Cancer.
Acronym: ARTSCAN V
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Version 2 2018-10-10
Record Dates: First submitted 2019-02-01; First posted 2019-02-04 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Tonsil Cancer
Keywords: Tonsil Cancer; Early Tonsil Cancer; Radiotherapy; Photons; Protons; Acute Side Effects; Late Side Effects; Locoregional Control; Disease Free Survival; Quality of Life; Health Economic
MeSH Terms: conditions — Tonsillar Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy delivered with photons (Active Comparator)
  Interventions: Radiation: Radiotherapy
- Radiotherapy delivered with protons (Experimental)
  Interventions: Radiation: Radiotherapy

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy with either photons or protons.

SUMMARY:
In this trial, patients with early squamous cell carcinoma of the tonsil with clinical stage T1-2 (p16-positive or p16-negative) N0-1 (p16-positive)/N0-N2b (p16-negative) according to American Joint Committee on Cancer (AJCC) 8th edition, aimed for unimodal and ipsilateral treatment with radiotherapy with curative intent will be included. The patients will be randomized to in a 1:1 ratio to receive radiotherapy with either photons (conventional radiotherapy) versus radiotherapy with protons.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be at least 18 years old.
2. Histologically or cytologically confirmed, previously untreated squamous cell carcinoma of the tonsil T1-2 (p16-positive or p16-negative) N0-1 M0 (p16-positive)/N0-N2b M0 (p16-negative) according to AJCC 8th edition, aimed for unimodal and ipsilateral treatment with radiotherapy with curative intent. The treatment may be followed but not preceded by surgery, which would be as a salvage procedure and not part of the planned treatment. An excision of a lymph node, or a tonsillectomy for diagnostic purposes does not exclude the patient from participation.
3. World Health Organisation/Eastern Cooperative Oncology Group (WHO/ECOG) performance status 0-1.
4. The patient must be able to understand the information about the treatment and give a written informed consent.

Exclusion Criteria:

1. Patients judged to benefit from bilateral radiotherapy or concomitant chemotherapy
2. Concomitant or previous malignancies. Exceptions are adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, or in situ carcinoma of the cervix uteri with a follow-up time of at least 3 years, or other previous malignancy with a disease-free interval of at least 5 years.
3. Two or more synchronous primary cancers in the head and neck region at time of diagnosis
4. Previous surgery or radiotherapy in the head and neck region that may affect the study result, as judged by the investigator
5. Co-existing disease prejudicing survival (expected survival should be >2 years).
6. Psychiatric or addictive disorders or other medical conditions which in the view of the investigator might impair patient compliance
7. When dental fillings with amalgam or metal are present close to the tumour area it must be considered if this may affect radiotherapy before inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Acute side effects. | From the third week of radiotherapy, and then weekly during radiotherapy, which ends after 7 weeks.
  Locoregional side effects (mucositis, pain, dysphagia, skin reactions and other functional impairment) are monitored weekly according to a modified morbidity scoring scale based on Radiation Therapy Oncology Group/European Organisation for Research and Treatment of Cancer (RTOG/EORTC). Acute radiation morbidity scoring criteria and other side effects are graded according to (Common Toxicity Criteria for Adverse Events (CTCAE) v4.0
Late side effects. | At 2-3 months after completed radiotherapy, then every 3 month for 2 years, and then every 6 month until 5 years.
  Locoregional side effects (mucositis, pain, dysphagia, skin reactions and other functional impairment) are monitored according to a modified morbidity scoring scale based on Radiation Therapy Oncology Group/European Organisation for Research and Treatment of Cancer (RTOG/EORTC). Late radiation morbidity scoring criteria and other side effects are graded according to Common Toxicity Criteria for Adverse Events (CTCAE) v4.0.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Gebre-Medhin, MD, Principal Investigator — Lund University Hospiyal
Locations (12):
- Sweden (12):
  - Gävle Hospital, Gävle
  - Sahlgrenska University Hospital, Gothenburg
  - Jönköping Hospital, Jönköping
  - Karlstad Hospital, Karlstad
  - Linköping University Hospital, Linköping
  - Lund University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - University Hospital, Umeå
  - Scandion clinic, Uppsala
  - Uppsala Accademical Hospital, Uppsala
  - Västmanlands Hospital, Västerås